CLINICAL TRIAL: NCT06967415
Title: Comparison of Pain, Central Sensitisation, Functional Status and Quality of Life According to Stenosis Degree in Individuals With Chronic Neck Pain
Brief Title: Comparison of Pain, Sensitisation, Function and Quality of Life According to Stenosis Degree in Chronic Neck Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Democracy University (Other)
Responsible Party: Principal Investigator, Ferruh Taşpınar, Prof. Dr., Izmir Democracy University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Central Sensitisation-35
Record Dates: First submitted 2025-04-22; First posted 2025-05-13 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Central Sensitisation; Cervical Spine Stenosis
Keywords: chronic neck pain
MeSH Terms: interventions — Central Nervous System Sensitization; Functional Status; Quality of Life

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- degree of cervical stenosis 0 (Other): Patients with a stenosis grade of 0 according to the Kang grading system in MRI imaging
  Interventions: Other: Pain, central sensitization,functional status and quality of life.
- degree of cervical stenosis 1 (Other): Patients with a stenosis grade of 1 according to the Kang grading system in MRI imaging
  Interventions: Other: Pain, central sensitization,functional status and quality of life.
- degree of cervical stenosis 2 (Other): Patients with a stenosis grade of 2 according to the Kang grading system in MRI imaging
  Interventions: Other: Pain, central sensitization,functional status and quality of life.
- degree of cervical stenosis 3 (Other): Patients with a stenosis grade of 3 according to the Kang grading system in MRI imaging
  Interventions: Other: Pain, central sensitization,functional status and quality of life.

INTERVENTIONS:
Other: Pain, central sensitization,functional status and quality of life. — The patients' pain status, central sensitization functional status, and quality of life will be evaluated according to their stenosis grade.

SUMMARY:
The cervical spine is a structure that bears the weight of the head and has important functions, but is susceptible to mechanical stress and degenerative processes. Cervical stenosis can lead to compression of the nerve roots as a result of narrowing of the spinal canal and symptoms such as pain, numbness and weakness. Central sensitisation (CS) causes even innocuous stimuli to cause pain due to hypersensitivity of the central nervous system and negatively affects the quality of life by increasing pain intensity in individuals with chronic neck pain. Progression of cervical stenosis can lead to symptoms such as walking difficulties, loss of balance and loss of proprioception. Furthermore, CS causes patients to avoid physical activity, increasing muscle weakness and pain, which further reduces quality of life. For this reason, our study will be carried out to determine the effect of cervical stenosis on patients with neck pain whom applied to Izmir Democracy University Physical Medicine and Rehabilitation outpatient clinic and had cervical MRI. Participants' pain status, central sensitisation, sensory loss, range of motion and proprioception will be recorded. Pressure pain threshold will be measured with algometer, sensory loss will be examined with Semmes-Weinstein Monofilament (SWM) Test, joint movements and proprioception will be evaluated with Pa CROM Basic device. In addition, the effects of cervical stenosis on functional status and quality of life will be measured by questionnaires. The data obtained will be compared and analysed with appropriate statistical methods. This study is aimed to contribute to the development of treatment methods and improvement of patient care, and will provide important information in terms of pain management and improvement of quality of life.

DETAILED DESCRIPTION:
The cervical spine is a critical structure that carries the entire weight of the head and protects the spinal cord, nerve roots and vertebral arteries. Since it is the most mobile part of the spine, it is the most exposed to mechanical stress, degenerative changes and trauma. Degenerative processes occurring in the cervical spine lead to conditions such as cervical spondylosis, cervical degenerative disc disease/disc herniation and cervical spondylotic myopathy, causing narrowing of the cervical spinal canal. A narrower than normal cervical spinal canal is defined as cervical spinal stenosis. In a study by Melancia et al., the researchers reported thatthe incidence of spinal stenosis is high in individuals aged 65 years and over, and that this condition may lead to symptoms such as pain, numbness, weakness, motor and sensory disorders as a result of compression of nerve roots.Neck pain is one of the most common musculoskeletal pathologies today. Global surveys show that a large proportion of the population experiences neck pain at some point in their lives. It is estimated that 50-85% of individuals with this condition will experience chronic pain within five years. Monticone et al. found that chronic neck pain has negative effects on quality of life as well as affecting activities of daily living. Chronic neck pain not only negatively affects the quality of life of individuals, but also imposes a serious burden on the health system.Neck pain is divided into different categories depending on its duration. If the pain persists for less than 6 weeks, it is considered acute neck pain. When the duration of pain is less than three months, it is classified as subacute neck pain, and when it lasts between three and six months, it is classified as chronic neck pain.There are many risk factors and causes that can lead to neck pain, such as poor posture, female gender and old age.Neck pain is a multifactorial condition with a variety of symptoms including decreased range of motion, asthenia, hyperalgesia and tension in superficial and deep neck muscles. With prolonged persistence of pain, some structural and sensory changes may occur in the central nervous system (CNS). These changes lead to increased stimulation of nociceptors and create an environment for the development of central sensitisation (CS). The International Association for the Study of Pain (IASP) defines central sensitisation (CS) as 'increased sensitivity of nociceptive neurons in the central nervous system to normal or subthreshold afferent inputs.Central sensitisation is a condition that occurs when pain transmission pathways are subjected to hypersensitivity. This process leads to an exaggerated perception of painful stimuli (hyperalgesia) and the perception of even harmless stimuli as pain (allodynia). However, central sensitisation plays a critical role in the development of reflected pain and hyperalgesia in multiple spinal segments. This mechanism triggers over-activation of the central nervous system, making individuals' pain experiences more intense. In this context, understanding central sensitisation is crucial for the development of chronic pain treatment strategies. Central sensitisation contributes tounderstand why individuals with musculoskeletal disorders experience pain, disability and other symptoms even in the absence of obvious nociceptive stimulation or tissue damage and in many diseases associated with chronic pain.While the existence of central sensitisation in chronic neck pain was the subject of debate in a study by Malfliet et al. in 2020, Roldán-Jiménez et al. observed that central sensitisation has a significant effect in different pain populations. The researchers found that central sensitisation is common especially among individuals with low back and neck pain.In a study conducted by Abdon et al. in 2024, indicated thatcentral sensitisation (CS) was more common in female individuals with chronic neck pain compared to male individuals with chronic neck pain. The symptoms associated with central sensitisation (CS) can increase the burden on health by complicating the treatment of patients and are therefore of great clinical importance. Studies have shown that patients with SS experience higher pain intensity, longer duration of pain, increased disability and decreased quality of life. The decline in functional status of individuals becomes more pronounced with increasing severity of CS.Although pain, functional status and quality of life are often assessed in individuals with cervical stenosis, there is a significant gap in the literature regarding the role of central sensitisation in these patients. Central sensitisation refers to an increased sensitivity of the central nervous system to pain and is known to be a pathological mechanism associated with chronic pain. However, studies on the presence and effects of central sensitisation in degenerative spine diseases such as cervical stenosis are limited. This deficiency represents a critical gap in the understanding of how to improve treatment strategies for patients with cervical stenosis. Evaluation of central sensitisation may provide a new perspective in the pain management of these patients and allow the development of more targeted treatment approaches. Therefore, our study was planned to examine the effects of the degree of cervical stenosis on central sensitisation, functional status and quality of life in individuals with chronic neck pain.

ELIGIBILITY:
Inclusion Criteria:

* Cases whose stenosis classification can be clearly determined on MRI
* Individuals with neck pain for at least 3 months

Exclusion Criteria:

* Individuals who did not agree to participate in the study
* Individuals undergoing cervical surgery
* Individuals with pain so severe that they cannot perform cervical movement
* Individuals with a diagnosis of vertigo
* Individuals with sudden hearing loss
* Individuals with additional neurological disorders
* Individuals with psychiatric and cognitive disorders that would prevent measurement in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-08-15 (Estimated)

PRIMARY OUTCOMES:
The assessment of pain. | Immediately after the stenosis grade is determined through MRI
  A Visual Analog Scale (VAS) will be used for pain assessment. The scale is 100 mm in length, with the words "no pain" and "the worst imaginable pain" fixed at the left and right ends. Individuals are asked to draw a vertical mark along the horizontal line that best represents their pain level. VAS is a widely used assessment method with good reliability and validity.
Central Sensitization Inventory (CSI) | Immediately after the stenosis grade is determined through MRI
  The Central Sensitization Inventory (CSI) will be used to assess central sensitization. This scale consists of a total of 25 items related to central sensitization symptoms, and participants are asked to mark a response ranging from "always" (four points) to "never" (zero points) for each item. The total score obtained from the scale ranges from 0 to 100, with a score of 40 or higher indicating the presence of central sensitization.
Pressure Pain Threshold (PPT) Measurement | Immediately after the stenosis grade is determined through MRI
  Pressure pain threshold measurement is a method performed using an algometer. In this method, the tip of the device is placed perpendicular to the area to be measured, and pressure is gradually increased. Measurements will be made bilaterally, and the areas to be measured include the Upper Trapezius muscle, Sternocleidomastoid muscle, and Cervical Erector Spinae muscle. The first pressure value at which the patient feels pain is recorded in kg/cm². This method is considered more economical and reliable compared to quantitative sensory tests.
Semmes-Weinstein Monofilament (SWM) Test | Immediately after the stenosis grade is determined through MRI
  The Semmes-weinstein monofilament test is one of the aesthesiometry tests used to evaluate tactile sensation in the clinical setting. It is tested with nylon monofilaments of approximately 38mm and varying diameters. The person is prevented from seeing the evaluation area and the person is explained how the test will be performed. In the area where the monofilament will be applied, pressure is applied to the skin in a perpendicular position (90⁰C angle) until the monofilament bulges. It is kept for 1.5 seconds in each region and the monofilament is removed from the skin after it is restored. The individual is asked to indicate 'yes' when he/she feels the stimulus on the skin. A maximum of 3 times stimulus is given in monofilaments from 1,65 to 4,08. For monofilaments from 4.17 to 6.65, 1 stimulus is given. If there is no response to the stimulus, the next filament is selected.
Copenhagen Neck Functional Disability Scale | Immediately after the stenosis grade is determined through MRI
  The scale, consisting of 15 items, measures the effects of neck pain (Jordan et al., 1998). In the scoring of the scale, points ranging from 0 to 2 are given based on the responses "Yes," "No," and "Sometimes." The maximum score that can be obtained from the scale is 30 points.
Assessment of Normal Joint Range of Motion | Immediately after the stenosis grade is determined through MRI
  Cervical region normal joint range of motion (ROM) will be assessed using the Pa Crom Basic - Cervical Range Of Motion (CROM) device. The CROM device is highly reliable for evaluating cervical joint range of motion. The device will be securely fixed to the patient's head using Velcro. Patients will be seated on a chair with their feet flat on the ground. The dial on the CROM will be set to the 0 position in the plane of the movement to be measured, and the correct movement technique will be taught to the patients. The patient will be asked to actively perform flexion, extension, right-left rotation, and right-left lateral flexion movements. Each movement will be repeated three times, and passive joint range of motion will be assessed. The average of the test values will be recorded.
Proprioceptive Sensory Assessment | Immediately after the stenosis grade is determined through MRI
  It will be assessed using the CROM device. Repositioning to a neutral head position (Joint Position Error - EPH) Repositioning the head to a predetermined reference point (Head Repositioning Accuracy - BYPD). For the BYPD test, the patient is asked to move the head to the target position. Deviations of 3-4 degrees from the target point indicate impaired joint position sense. patient sits upright. The CROM device is placed on the patient's head with velcro. Deviations in the dials on the CROM device are recorded. For the BYPD test, half of the measured maximum active range of motion is set as the target position. With the patient's eyes closed, the head is slowly moved to the target position and perceived. Then the head is moved in the opposite direction and the patient actively brings the head to this position. Measurements are made 3 times and the average deviation is recorded. Measurements are made for flexion, extension, right-left rotation and right-left lateral flexion.
Quality of Life Assessment | Immediately after the stenosis grade is determined through MRI
  The Short Form-36 (SF-36) will be used. This questionnaire examines 8 dimensions of health with 36 items. These dimensions include social functioning, physical functioning, physical role limitations, energy, mental health, emotional role limitations, general health perception, and pain. When there are no limitations or disabilities, the highest possible score of 100 is obtained. Each dimension is evaluated independently, and a higher score indicates a higher quality of life for that dimension.

CONTACTS AND LOCATIONS:
Overall Officials: Onur Engin, Assist Prof, Principal Investigator — Izmir Democracy University
Locations (1):
- Izmir Democracy University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No